CLINICAL TRIAL: NCT02055456
Title: Male Hormones for Telomere Related Diseases
Brief Title: Nandrolone Decanoate in the Treatment of Telomeropathies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Diego Villa Clé, MD, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-H-RTC-0002
Record Dates: First submitted 2014-02-03; First posted 2014-02-05 (Estimated); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Aplastic Anemia; Bone Marrow Failure Syndromes; Idiopathic Pulmonary Fibrosis; Telomere Shortening
Keywords: Hormones; Androgens; Aplastic Anemia; Bone Marrow Failure Syndromes; Idiopathic Pulmonary Fibrosis; Telomere; Telomere Shortening
MeSH Terms: conditions — Anemia, Aplastic; Bone Marrow Failure Disorders; Idiopathic Pulmonary Fibrosis | interventions — Nandrolone Decanoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nandrolone Decanoate (Experimental): Nandrolone Decanoate intramuscularly administered, every two weeks, 5 mg/kg/dose
  Interventions: Drug: Nandrolone Decanoate

INTERVENTIONS:
Drug: Nandrolone Decanoate

SUMMARY:
Decrease in blood cell counts due to deficient bone marrow function, called bone marrow failure, as well as some lung diseases, called idiopathic pulmonary fibrosis, can be caused by genetic defects in telomere biology genes, eventually causing telomere erosion. These disorders are collectively termed "telomeropathies".

There is evidence that male hormones may improve blood cell counts in marrow failure, and these hormones are able to stimulate telomerase function in hematopoietic cells in vitro. We propose this study to the use of male hormone in patients with aplastic anemia and pulmonary fibrosis associated with defects in telomeres.

DETAILED DESCRIPTION:
Telomeres are repeated nucleotide sequences of non-coding DNA at the ends of chromosomes that have protective functions and avoid chromosomes recombinations and fusions.

Loss-of-function mutations in genes of the telomerase complex, a enzyme responsible for maintaining telomere length, has been associated with bone marrow failures, notedly mutations in DKC1 gene, detected in a rare inherited form of marrow aplasia, called dyskeratosis congenita. These findings implicated telomerase dysfunction and shortening telomere length in failed hematopoiesis.

In family members of probands with aplastic anemia, marrow aplasia and telomerase mutations also have been observed and associated to varying degrees of cytopenias, IPF and/or cirrhosis. Moreover, patients with varying degrees of cytopenias, with significant family history for cytopenias, IPF and/or cirrhosis, have been identified with very short telomeres and some mutations in telomerase complex genes. Additionally, telomere length has been associated with human cancer.

In vitro studies suggest that telomere length could be modulated with sex hormones. Normal lymphocytes and human bone marrow progenitor cells exposed to androgens increased telomerase activity in vitro, and in individuals with telomerase mutations (TERT) androgens increased telomerase activity.This could be the explanation for the hematologic improvement observed in some aplastic anemia patients treated over 40 years ago with male hormones.

Therefore, we hypothesize that androgens therapy might modulate telomere attrition in vivo and ameliorate progression or reverse the clinical consequences of shortening telomere length, and we propose androgens therapy in patients with cytopenias and/or IPF with a short age adjusted telomere length, with or without telomerase gene mutations.

The primary biologic endpoint will be the reduction of telomere attrition over time compared to known rates of telomere erosion in normal individuals and in those who carry mutation in the telomerase genes. Secondary endpoints will be tolerability of nandrolone decanoate over two years, improvement in blood counts and/or pulmonary function.

ELIGIBILITY:
Inclusion Criteria:

* Peripheral blood leukocytes telomeres short for age, below the first percentile of a curve based on 500 healthy individuals between 0 and 100 years, with or without a telomerase gene mutation.

AND

* One or more of the following cytopenias:

Anemia (symptoms of anemia with hemoglobin <9.5 g/dL, or need for transfusion > 2 units of packed red blood cells/month for at least two months, or absolute reticulocytes count <60.000/μL).

Thrombocytopenia (platelets counts <30.000/μL or <50.000/μL associated with bleeding, or megakaryocytes reduction in the bone marrow).

Neutropenia (absolute neutrophil counts <1.000/μL).

OR

* Idiopathic pulmonary fibrosis diagnosed according to the American Thoracic Society (ATS) criteria.

Exclusion Criteria:

* Terminal disease or liver disease, renal, cardiac, neurological, infectious or concomitant metabolic state whose gravity prevents the ability of the patient to tolerate the treatment protocol, or probable death within 30 days.
* People with cancer who are undergoing chemotherapy.
* Pregnancy, or desire to not prevent pregnancy in childbearing age.
* Aplastic Anemia patients with indication for bone marrow transplantation and matched donor.

Ages: 2 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Reduction in telomere attrition | 2 years
  The biologic endpoint is reduction in telomere attrition rate yearly compared to known rates of telomere erosion in normal individuals and in those who carry mutation in the telomerase genes

SECONDARY OUTCOMES:
Hematologic response | 2 years
  The hematologic response will be determined by one or more of the following:
  1. absolute neutrophil counts (increase of more than 500/μL above initial value)
  2. platelets (increase of more than 20.000/μL above initial value)
  3. Hemoglobin:
     * Increase in hemoglobin of more than 1.5 g/dL above initial value OR
     * Transfusion independence in transfusion-dependent patients (more than 2 months without transfusion) OR
     * Reduction of the transfusion needs in more than 50%
Clonal evolution | 2 years
  Number of participants that evolute to myelodysplasia or acute leukemia.
Improvement in lung function | 2 years
  The pulmonary response will be determined by the presence of one or more of the following:
  1. Improvement of dyspnea severity, objectively evaluated by "Baseline Dyspnea Index";
  2. forced vital capacity (10% absolute increase)
  3. Diffusion of carbon monoxide (DLCO) corrected for hemoglobin (15% increase)
  4. No worsening of pulmonary fibrosis and reduction of assessed ground-glass opacities in computed tomography of the chest
Survival | 2 years
Safety | 2 years
  Number of participants with adverse effects attributed to the use of nandrolone decanoate during the 24 months treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo T Calado, MD, PhD, Study Chair — Ribeirao Preto School of Medicine at University of Sao Paulo; Diego V Clé, MD, Principal Investigator — Ribeirao Preto School of Medicine at University of Sao Paulo; Ana Beatriz Hortense, MD, Principal Investigator — Ribeirao Preto School of Medicine at University of Sao Paulo; José Antonio Baddini Martinez, MD, PhD, Study Chair — Ribeirao Preto School of Medicine at University of Sao Paulo
Locations (1):
- Ribeirao Preto School of Medicine, University of Sao Paulo, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Background] Young NS, Calado RT, Scheinberg P. Current concepts in the pathophysiology and treatment of aplastic anemia. Blood. 2006 Oct 15;108(8):2509-19. doi: 10.1182/blood-2006-03-010777. Epub 2006 Jun 15. PMID 16778145
- [Background] Calado RT, Young NS. Telomere maintenance and human bone marrow failure. Blood. 2008 May 1;111(9):4446-55. doi: 10.1182/blood-2007-08-019729. Epub 2008 Jan 31. PMID 18239083
- [Background] Yamaguchi H, Calado RT, Ly H, Kajigaya S, Baerlocher GM, Chanock SJ, Lansdorp PM, Young NS. Mutations in TERT, the gene for telomerase reverse transcriptase, in aplastic anemia. N Engl J Med. 2005 Apr 7;352(14):1413-24. doi: 10.1056/NEJMoa042980. PMID 15814878
- [Background] Calado RT, Yewdell WT, Wilkerson KL, Regal JA, Kajigaya S, Stratakis CA, Young NS. Sex hormones, acting on the TERT gene, increase telomerase activity in human primary hematopoietic cells. Blood. 2009 Sep 10;114(11):2236-43. doi: 10.1182/blood-2008-09-178871. Epub 2009 Jun 26. PMID 19561322
- [Background] Calado RT, Young NS. Telomere diseases. N Engl J Med. 2009 Dec 10;361(24):2353-65. doi: 10.1056/NEJMra0903373. No abstract available. PMID 20007561
- [Background] Ziegler P, Schrezenmeier H, Akkad J, Brassat U, Vankann L, Panse J, Wilop S, Balabanov S, Schwarz K, Martens UM, Brummendorf TH. Telomere elongation and clinical response to androgen treatment in a patient with aplastic anemia and a heterozygous hTERT gene mutation. Ann Hematol. 2012 Jul;91(7):1115-20. doi: 10.1007/s00277-012-1454-x. Epub 2012 Apr 4. PMID 22476886
- [Derived] Cle DV, Catto LFB, Gutierrez-Rodrigues F, Donaires FS, Pinto AL, Santana BA, Darrigo LG, Valera ET, Koenigkam-Santos M, Baddini-Martinez J, Young NS, Martinez EZ, Calado RT. Effects of nandrolone decanoate on telomere length and clinical outcome in patients with telomeropathies: a prospective trial. Haematologica. 2023 May 1;108(5):1300-1312. doi: 10.3324/haematol.2022.281808. PMID 36579443